CLINICAL TRIAL: NCT04146662
Title: The Performance of Faecal Immunochemical Test and Urinary Volatile Compounds in the Detection of Colorectal Adenomas and Their Role in Polyp Surveillance
Brief Title: Faecal Immunochemical Test and Urine Volatile Compounds in Adenoma Detection
Acronym: FASt
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RA433019
Record Dates: First submitted 2019-10-10; First posted 2019-10-31 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine, Stool, and Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Faecal immunochemical test — Faecal immunochemical test (FIT) and urine volatile organic compounds (VOC) analysis.
  Other Names: Urine volatile organic compounds

SUMMARY:
Bowel cancer can arise from polyps, which can become cancerous. Polyps are little outgrowths within the lining of the bowel (similar to skin warts). Depending on their size and their potential to become cancerous, they can cause bleeding. However, it is not known which polyps harbour cancerous potential. Therefore, at present all patients undergo a colonoscopy (camera examination of the large bowel) in order to identify and remove any polyps. However, not all patients who undergo a colonoscopy will have polyps. Moreover, colonoscopies are invasive and disruptive to patients, as they require bowel preparation. The aim of this study is to evaluate non-invasive stool and urine tests to identify patients who are at risk of polyps and if the polyps have the potential to become cancerous. This in turn, will significantly reduce the number of 'unnecessary' polyp surveillance colonoscopies with resultant benefits to both patients and the National Health Service (NHS).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are on a polyp surveillance programme and will be undergoing colonoscopy examination for polyp surveillance OR Patients who will be undergoing elective polypectomy through specialised polyp multi-disciplinary meetings.

Exclusion Criteria:

* Participants who are unable to attend colonoscopy
* Under 18 years old
* Unable to provide informed consent for themselves to take part in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over 18 years who are known to have colorectal polyps and on polyp surveillance programme
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Faecal immunochemical test and urine volatile markers to detect colorectal adenomas | Through study completion, an average of 2 years
  To determine the sensitivity of Faecal immunochemical test and urine volatile markers to detect colorectal adenomas - individually and in combination, in comparison to colonoscopy results (histology findings).

SECONDARY OUTCOMES:
Sensitivity of Faecal immunochemical test and urine volatile markers for all adenomas and high-grade adenomas | Through study completion, an average of 2 years
  To determine the specificity and receiver operator curve for Faecal immunochemical test and urine volatile markers for all adenomas and high-grade adenomas.
Positivity threshold for Faecal immunochemical test and urine volatile markers | Through study completion, an average of 2 years
  To determine the positivity threshold for FIT and urine VOC for detection of adenomas, comparing all adenomas vs high grade adenomas.
Volatile chemicals in urine in those with adenomas | Through study completion, an average of 2 years
  To identify the specific volatile chemicals that are consistently present in those with adenomas.
To determine the sensitivity of blood markers for the detection of colorectal adenomas | Through study completion, an average of 2 years
  To determine the sensitivity of blood markers e.g. Septin 9 for the detection of colorectal adenomas

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Coventry & Warwickshire NHS Trust, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided